CLINICAL TRIAL: NCT05280704
Title: Traditional Dorsal Digital Block Vs Volar Subcutaneous Digital Block
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Slow accrual and other non-safety related issues
Sponsor: University of Arkansas (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 274026
Record Dates: First submitted 2022-03-04; First posted 2022-03-15 (Actual); Last update posted 2024-11-18 (Actual); Status verified 2024-11

CONDITIONS: Hand Injuries
Keywords: digital block
MeSH Terms: conditions — Hand Injuries | interventions — Lidocaine; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: Our study design is a two-period cross-over design with four groups defined by order of treatment, in which each subject will experience both injection techniques, one to each hand.
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Each participant will collect two syringes with a code indicting the order and technique of injection. The contents of the syringe (lidocaine vs normal saline) will not be known by the care provider, outcomes assessor or participant.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- V1 Lidocaine, D2 Saline (Other): Will undergo volar technique 1st with 4 mL of 1% lidocaine and then dorsal technique 2nd with 4 mL of 0.9% sterile saline. This is a 1-time dose.
  Interventions: Procedure: Volar digital block with lidocaine; Procedure: Dorsal digital block with saline
- V1 Saline, D2 Lidocaine (Other): Will undergo volar technique 1st with 4 mL of 0.9% sterile saline and then dorsal technique 2nd with 4 mL of 1% lidocaine. This is a 1-time dose.
  Interventions: Procedure: Volar digital block with saline; Procedure: Dorsal digital block with lidocaine
- D1 Lidocaine, V2 Saline (Other): Will undergo dorsal technique first with 4 mL of 1% lidocaine and then volar technique second with 0.9% sterile saline. This is a 1-time dose.
  Interventions: Procedure: Volar digital block with saline; Procedure: Dorsal digital block with lidocaine
- D1 Saline, V2 Lidocaine (Other): Will undergo dorsal technique 1st with 4 mL of 0.9% sterile saline and then volar technique 2nd with 4 mL of 1% lidocaine. This is a 1-time dose.
  Interventions: Procedure: Volar digital block with lidocaine; Procedure: Dorsal digital block with saline

INTERVENTIONS:
Procedure: Volar digital block with lidocaine — Volar digital block with lidocaine
  Arms: D1 Saline, V2 Lidocaine; V1 Lidocaine, D2 Saline
Procedure: Volar digital block with saline — Volar digital block with saline
  Arms: D1 Lidocaine, V2 Saline; V1 Saline, D2 Lidocaine
Procedure: Dorsal digital block with lidocaine — Dorsal digital block with lidocaine
  Arms: D1 Lidocaine, V2 Saline; V1 Saline, D2 Lidocaine
Procedure: Dorsal digital block with saline — Dorsal digital block with saline
  Arms: D1 Saline, V2 Lidocaine; V1 Lidocaine, D2 Saline

SUMMARY:
This is a prospective, randomized, double-blinded controlled trial comparing two different techniques for digital blocks. Participants will be physicians who perform digital blocks as part of their everyday duty. Each participant will undergo two digital blocks and will have the opportunity to perform a digital block on another participant.

This study follows a two-period cross-over design with four groups that are defined by the sequence of treatments within each group. Participants will receive two digital blocks, one using the traditional dorsal technique and one using the volar technique. Of the two injections, one of the syringes will contain 1% lidocaine without epinephrine and the other will contain sterile normal saline. The injections will be to the index finger on each hand. The hand injected first will be up to the participant. The order in which the dorsal technique versus the volar technique is performed will be randomized. Participants will not be told one of the syringes contains normal saline. Injection pain will be measured by visual analog score and recorded after each injection. Sensation in each of the 12 zones of the finger will be recorded at each minute mark until loss of sensation in all 12 zones is achieved or 15 minutes has passed, whichever comes first.

DETAILED DESCRIPTION:
This is a prospective, randomized, double-blinded controlled trial comparing two different techniques for digital blocks. Participants will be physicians who perform digital blocks as part of their everyday duty. Each participant will undergo two digital blocks and will have the opportunity to perform a digital block on another participant.

This study follows a two-period cross-over design with four groups that are defined by the sequence of treatments within each group. Participants will receive two digital blocks, one using the traditional dorsal technique and one using the volar technique. Of the two injections, one of the syringes will contain 1% lidocaine without epinephrine and the other will contain sterile normal saline. The injections will be to the index finger on each hand. The hand injected first will be up to the participant. The order in which the dorsal technique versus the volar technique is performed will be randomized. Participants will not be told one of the syringes contains normal saline. Injection pain will be measured by visual analog score and recorded after each injection. Sensation in each of the 12 zones of the finger described by Cummings et al will be recorded at each minute mark until loss of sensation in all 12 zones is achieved or 15 minutes has passed, whichever comes first.

Set Up Prior to Study Performance Four-digit codes will be created for all participants. The 4-digit codes will be randomly assigned to a treatment group, A, B, C and D. Group A will undergo the volar technique first with lidocaine (V1) and then the dorsal technique second with sterile saline (D2). Group B will undergo the volar technique first with sterile saline and then undergo the second injection with the dorsal technique with lidocaine. Group C will undergo the dorsal technique first with lidocaine (D1) and then the volar technique second with sterile saline (V2). Group D will undergo the dorsal technique first with sterile saline followed by the volar technique second with lidocaine. Two syringes will be prepared for each 4-digit code, one with 4 mL of 1% lidocaine and 4 mL of sterile normal saline. They will be labelled with the four-digit code and a separate letter-digit code. The letter-digit code will contain one letter, either V or D, and one number, 1 or 2. The letter corresponds to the technique used to perform the injection (V for volar technique, D for traditional dorsal technique). The number corresponds to the order to which the syringe is to be used, first or second. Figure 1 shows a typical example of how a syringe will be labelled. In this example, participant 4883 in Group A would receive a syringe of lidocaine labelled 4883 V1 and a syringe of saline labelled 4883 D2. Each syringe will also be marked with an * indicating lidocaine and a # indicating sterile saline. This is added to the syringes to immediately determine the syringe contents in case of adverse reaction. The meaning of the * and # will not be shared with participants but will be known to all members of the study team.

Date of Study

An anonymous survey will be given to all participants with three questions:

1. Which technique do participants use for digital blocks?
2. How many mLs of lidocaine do participants use for digital block of one finger?
3. What specialty of medicine do participants practice? A ten-minute instructional demonstration will be performed demonstrating the volar injection technique and the traditional dorsal digital block technique as well as explaining the pain visual analog scale, the 12 zones of the finger, and how to record the data.

Participants will collect their two syringes with the same four-digit code. They will not be told that one syringe contains normal saline. Participants will then pair into groups of three. Within a group of three, each participant will be assigned the role of subject, injector, or recorder. The recorder will record the 4- digit number code at the top of the data sheet for the subject prior to injection. The injector will prep the base of the subject's index finger and perform the digital block in a sterile fashion using the technique indicated by letter on the syringe labeled 1. The recorder will start the timer. Pain on injection using the Visual Analog Score (VAS) will be recorded. Pinprick sensation will be tested in all 12 zones of the finger and recorded by the recorder at each minute mark up to 15 minutes or loss of sensation in all 12 zones, whichever comes first. The injector will then prep the base of the index finger on the subject's other hand and proceed with the second digital block using the technique corresponding to the letter on the syringe labelled 2. Again, pain on injection using the VAS will be recorded, pinprick sensation will be tested in all 12 zones of the finger and recorded by the recorder at each minute mark up to 15 minutes or loss of sensation in all 12 zones of the finger. Subject will then record which injection they prefer based on the pain on injection, not on the efficacy of technique at achieving loss of sensation. The participants will switch, so that the injector will become the subject, the recorder will become the injector, the subject will become the recorder, and the above-described procedure will be repeated. Then the participants will switch once more, and same procedure will be conducted a third and final time. If the injector in the final round has an insensate index finger, then an injector from another group with a sensate digit will perform the injections.

Participants may withdraw from the study at any time without prejudice to their training. Under certain circumstances the researchers may terminate the participant's participation in the study if: the participant is found to meet exclusion criteria, it is not in the participant's best interest to continue, or the study is stopped for any reason.

ELIGIBILITY:
Inclusion Criteria:

* Physicians over the age of 18 who regularly perform digital blocks as part of their duty, including those who specialize in Orthopaedic Surgery, Pediatrics, Family Medicine and Emergency Medicine.

Exclusion Criteria:

* Participants with absence of an index finger on either side
* Pregnancy
* Neuropathy
* Hematologic disease
* Peripheral vascular disease
* Participants with a history of adverse reactions to lidocaine

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2023-09-20 (Actual); Primary Completion 2023-09-20 (Actual); Study Completion 2023-09-20 (Actual)

PRIMARY OUTCOMES:
Injection Pain | Immediately upon injection
  The primary outcome is injection pain as measured by the visual analog score (VAS). The VAS for pain is a straight line with one end meaning no pain and the other end meaning the worst pain imaginable. A patient indicates a point on the line that matches the amount of pain he or she feels. Data for this outcome will be analyzed using mixed-models ANOVA with Subject as the random effect. The fixed effects in the ANOVA model will be the Technique main effect, the Agent main effect, the Technique-x-Agent interaction, and the Order main effect. Because each subject's two treatments will be administered to opposite hands, there should be no carryover effects, and the ANOVA model accordingly will not include Order interactions with Technique or Agent.

SECONDARY OUTCOMES:
Efficacy of Desensitization | Pinprick sensation will be tested in all 12 zones of the finger and recorded by the recorder at each minute mark up to 15 minutes or loss of sensation in all 12 zones, whichever comes first.
  Time to loss of sensation in all 12 finger zones will be right-censored at the 15-minute mark, graphed as Kaplan-Meier curves, and, depending on distributional characteristics, compared for a Volar-versus-Dorsal difference using either the log-rank test or the Gehan-Wilcoxon test at P<0.05 (2-sided).

CONTACTS AND LOCATIONS:
Overall Officials: Sean Morell, MD, Principal Investigator — University of Arkansas
Locations (1):
- University of Arkansas for Medical Sciences, Little Rock, Arkansas, United States

IPD SHARING:
Plan to Share IPD: No
Upon enrollment, each study participant will be assigned a unique identifying code (Participant ID), which will be used in place of their name on study documents to create a de-identified dataset. The key to this code will be kept separately from study data and will be stored in a locked file in Orthopedics office at UAMS. Only study personnel will have access to the code and any information that identifies the participant in this study. Once accepted for publication, the documents containing the unique study codes associated with the subjects' names will be destroyed.

REFERENCES:
- [Background] Ito N, Umazume M, Ojima Y, Shibata D, Ida Y, Komiya T, Matsumura H. Comparison of traditional two-injection dorsal digital block versus transthecal and subcutaneous single-injection digital block: A systematic review and meta-analysis. Hand Surg Rehabil. 2021 Sep;40(4):369-376. doi: 10.1016/j.hansur.2021.04.004. Epub 2021 Apr 23. PMID 33895422
- [Background] Whetzel TP, Mabourakh S, Barkhordar R. Modified transthecal digital block. J Hand Surg Am. 1997 Mar;22(2):361-3. doi: 10.1016/S0363-5023(97)80179-7. No abstract available. PMID 9195442
- [Background] Cummings AJ, Tisol WB, Meyer LE. Modified transthecal digital block versus traditional digital block for anesthesia of the finger. J Hand Surg Am. 2004 Jan;29(1):44-8. doi: 10.1016/j.jhsa.2003.09.018. PMID 14751102
- [Background] Braun H, Harris ML. Operations on the extremities. In: Local Anesthesia: It's Scientific Basis and Practical Use. 2nd ed. Lea & Febiger; 1924:366-367.
- [Background] Williams JG, Lalonde DH. Randomized comparison of the single-injection volar subcutaneous block and the two-injection dorsal block for digital anesthesia. Plast Reconstr Surg. 2006 Oct;118(5):1195-1200. doi: 10.1097/01.prs.0000237016.00941.96. PMID 17016190
- [Background] Harbison S. "Transthecal digital block: flexor tendon sheath used for anaesthetic infusion". J Hand Surg Am. 1991 Sep;16(5):957. doi: 10.1016/s0363-5023(10)80172-8. No abstract available. PMID 1940182
- [Background] Yin ZG, Zhang JB, Kan SL, Wang P. A comparison of traditional digital blocks and single subcutaneous palmar injection blocks at the base of the finger and a meta-analysis of the digital block trials. J Hand Surg Br. 2006 Oct;31(5):547-55. doi: 10.1016/j.jhsb.2006.06.001. Epub 2006 Aug 22. PMID 16930788
- [Background] Bashir MM, Khan FA, Afzal S, Khan BA. Comparison of traditional two injections dorsal digital block with volar block. J Coll Physicians Surg Pak. 2008 Dec;18(12):768-70. PMID 19032891
- [Background] Martin SP, Chu KH, Mahmoud I, Greenslade JH, Brown AF. Double-dorsal versus single-volar digital subcutaneous anaesthetic injection for finger injuries in the emergency department: A randomised controlled trial. Emerg Med Australas. 2016 Apr;28(2):193-8. doi: 10.1111/1742-6723.12559. Epub 2016 Mar 16. PMID 26991958
- [Background] Afridi RA, Masood T, Ahmed E, Obaidullah AM, Alvi HF. Comparison of the efficacy of single volar subcutaneous digital block and the dorsal two injections block. J Ayub Med Coll Abbottabad. 2014 Jan-Mar;26(1):88-91. PMID 25358227
- [Background] Okur OM, Sener A, Kavakli HS, Celik GK, Dogan NO, Icme F, Gunaydin GP. Two injection digital block versus single subcutaneous palmar injection block for finger lacerations. Eur J Trauma Emerg Surg. 2017 Dec;43(6):863-868. doi: 10.1007/s00068-016-0727-9. Epub 2016 Oct 5. PMID 27709248
- [Background] Cannon B, Chan L, Rowlinson JS, Baker M, Clancy M. Digital anaesthesia: one injection or two? Emerg Med J. 2010 Jul;27(7):533-6. doi: 10.1136/emj.2009.072850. Epub 2010 Apr 1. PMID 20360491